CLINICAL TRIAL: NCT07096232
Title: Orchestrated Multi Agent Artificial Intelligence (AI) Versus Consultant Ophthalmologist: Workflow Performance in Refractive Surgery and Keratoconus Diagnosis. Demonstrating Increased Diagnostic Accuracy (Automated Evaluation for Your Eye, AEYE).
Brief Title: AI-Orchestrated Workflow Versus Consultant Ophthalmologist for Refractive Surgery and Keratoconus Diagnosis (AEYE Trial)
Acronym: AEYE
Status: Enrolling by invitation | Type: Observational
Sponsor: Hazem Yassin Clinics (Other)
Collaborators: Ahmed I ElSayegh (Unknown)
Responsible Party: Principal Investigator, hatem ali, Doctor, Hazem Yassin Clinics
Other Study IDs: HYC-AI-RS-2025-01
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus; Refractive Surgery; Machine Learning; Artifical Intelligence; Diagnostic Accuracy; Clinical Decision Support; Ophthalmology
Keywords: Keratoconus; Corneal Diseases; Refractive Surgical Procedures; Anterior Eye Segment; Diagnostic Imaging; Artificial Intelligence; Diagnostic Techniques, Ophthalmological; Clinical Decision-Making; AI-Assisted Diagnosis
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with refractive errors or keratoconus assessed by agentic AI workflow and consultant review: This group includes all patients with refractive errors or keratoconus evaluated at our center during the study period. Each patient case undergoes comprehensive diagnostic assessment using both an orchestrated multi-agent artificial intelligence (AI) workflow (AEYE) and independent review by a consultant ophthalmologist. The AI workflow integrates multiple specialized AI agents to analyze clinical data, imaging studies, and relevant diagnostic metrics. Results from the AI system are compared to consultant assessments to evaluate concordance, diagnostic accuracy, and workflow efficiency. Both retrospective patient records and prospectively enrolled cases are included in this group.
  Interventions: Diagnostic Test: Multi-Agent AI Diagnostic Workflow (AEYE)

INTERVENTIONS:
Diagnostic Test: Multi-Agent AI Diagnostic Workflow (AEYE) — This intervention consists of an orchestrated diagnostic workflow utilizing multiple specialized artificial intelligence (AI) agents to analyze patient data and ophthalmic imaging for the diagnosis of refractive errors and keratoconus. The workflow, named Automated Evaluation for Your Eye (AEYE), integrates various AI modules designed for data extraction, image interpretation, and decision support. Each patient's clinical information, corneal topography, tomography, and other relevant imaging are processed sequentially through these AI agents, with results synthesized into a diagnostic recommendation. The system operates independently of clinician input, and outputs are blinded prior to comparison with consultant ophthalmologist assessments. The intervention is intended to assess diagnostic accuracy, efficiency, and concordance with expert clinical decision-making.
  Other Names: Automated Evaluation for Your Eye, AI Workflo; Artificial Intelligence assisted Diagnostic workflow for Keratoconus and Refractive Surgery Evaluation

SUMMARY:
Background and Rationale:

Laser vision correction procedures, such as LASIK (Laser-Assisted In Situ Keratomileusis), PRK (Photorefractive Keratectomy), and SMILE (Small Incision Lenticule Extraction), are highly effective but require careful preoperative screening to ensure safety. One of the most critical aspects of screening is identifying keratoconus and other corneal ectatic disorders-conditions that cause progressive thinning and bulging of the cornea, often contraindicating surgery. Early detection is essential to avoid vision-threatening complications.

Despite advanced corneal imaging tools such as Scheimpflug tomography and anterior segment optical coherence tomography (AS-OCT), accurate diagnosis-particularly in borderline or early-stage cases-remains challenging and subject to variability in human interpretation. Artificial intelligence (AI) offers the potential to improve diagnostic precision, reduce oversight, and standardize surgical planning.

Purpose of the Study:

This study evaluates the performance of AEYE (Automated Evaluation for Your Eye), a multi-agent AI system designed to support ophthalmologists in diagnosing keratoconus and determining refractive surgery eligibility. AEYE simulates the clinical workflow of an anterior segment specialist by orchestrating three specialized agents:

History & Risk Agent: Reviews patient history and extracts risk factors.

Imaging Agent: Analyzes corneal tomography, AS-OCT, and epithelial mapping scans.

Surgical Decision Agent: Integrates all findings, assigns a diagnosis, and recommends appropriate treatment options, including surgical eligibility or corneal cross-linking (CXL).

Study Design:

The study includes 50 real-world patient cases, both retrospective (from 2020 onward) and prospective, who were evaluated for refractive surgery or keratoconus. Each case is analyzed independently by AEYE and a consultant ophthalmologist (blinded to AI output), using the same multimodal clinical and imaging data. Diagnostic accuracy, agreement in surgical recommendations, and workflow efficiency are assessed.

Anticipated Impact:

By comparing AI-derived decisions with expert clinical judgment, this study aims to validate whether structured AI workflows like AEYE can serve as reliable, safe, and explainable decision support tools. If successful, AEYE may offer a scalable solution to reduce diagnostic variability and enhance the safety and consistency of refractive surgery screening.

DETAILED DESCRIPTION:
Technical Protocol Summary

This is a diagnostic performance study evaluating AEYE (Automated Evaluation for Your Eye), an orchestrated multi-agent artificial intelligence (AI) system designed to assist ophthalmologists in the screening and management of keratoconus and refractive surgery planning. AEYE combines large language models (LLMs) with deterministic code logic to replicate and support the clinical decision-making process typically performed by anterior segment specialists.

System Architecture and Workflow

AEYE is structured as a modular pipeline of three specialized agents, each focused on a distinct diagnostic task:

History and Risk Agent: Extracts structured data from unstructured clinical records, including demographics, ocular/systemic history, medication use, and risk factors relevant to keratoconus or refractive surgery eligibility.

Imaging Analysis Agent: Processes multimodal anterior segment imaging such as Scheimpflug-based tomography (e.g., Pentacam), anterior segment optical coherence tomography (AS-OCT), and epithelial thickness mapping. It standardizes key metrics like maximum keratometry (Kmax), thinnest corneal pachymetry, anterior/posterior elevation, Belin-Ambrósio Deviation Index (BAD-D), and Pachymetric Progression Index (PPI). Each eye and each imaging file is processed independently to avoid misattribution.

Surgical Decision Agent: Integrates the outputs of the previous agents to generate a final diagnosis, assign keratoconus staging (e.g., ABCD, Amsler-Krumeich classification), and recommend next steps, such as LASIK (Laser-Assisted In Situ Keratomileusis), PRK (Photorefractive Keratectomy), SMILE (Small Incision Lenticule Extraction), phakic intraocular lenses (ICL), or corneal collagen cross-linking (CXL). The output is a structured, auditable report.

All agents are controlled by a deterministic workflow using Python scripts for data merging, schema validation, and output formatting. Structured memory is maintained using JSON objects that store the full diagnostic context per patient. The system is designed to ensure reproducibility, reduce human variability, and support explainable clinical decision-making.

Study Workflow and Scope

Fifty real-world patient cases are included, comprising both retrospective records (from January 2020 onward) and newly enrolled prospective cases. Each case includes comprehensive clinical data and anterior segment imaging. AEYE analyzes the case and generates a structured report. Separately, an experienced ophthalmologist (blinded to the AI output) reviews the same data and records their clinical decisions.

Key metrics include:

Diagnostic accuracy of keratoconus detection. Agreement in surgical eligibility assessments. Efficiency of workflow execution. Variability in results across different LLMs used in agent roles. Cases with discordant results may undergo adjudication to establish a reference standard.

Innovation and Clinical Relevance.

AEYE represents a novel application of explainable AI in ophthalmology. Its multi-agent design reflects a divide-and-conquer strategy, reducing cognitive load on any single model while enforcing clinical safety through deterministic logic. The system supports scalability, modularity, and integration into electronic health record (EHR) systems. The study will help determine whether AEYE can function as a safe, consistent, and effective assistant in complex diagnostic pathways for corneal ectatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Refractive Error or Keratoconus:

   * Patients with a confirmed clinical diagnosis of refractive errors (myopia, hyperopia, or astigmatism) or keratoconus, as determined by a qualified ophthalmologist based on current diagnostic standards.
2. Availability of Complete Data:

   * Clinical records must include comprehensive demographic data, medical and ophthalmic history, refraction measurements, and high-quality corneal imaging (e.g., corneal topography, tomography, or OCT).
3. Eligible for Both AI and Consultant Review:

   * Patients must have data sets that allow both the multi-agent AI workflow (AEYE) and an independent consultant ophthalmologist to conduct a complete diagnostic assessment.
4. Consent:

   * For prospectively enrolled patients, written informed consent must be obtained prior to participation. For retrospective cases, waiver of consent may be granted according to local IRB/ethics committee policies.
5. No Restriction on Age or Sex:

   * There are no specific age or sex limitations for inclusion in this study. Pediatric and adult cases may be included if data are available and consent is appropriately obtained.

Clinical Documentation Requirements:

* Availability of complete ophthalmic records including:
* Uncorrected and best corrected visual acuity (UCVA, BCVA)
* Manifest refraction (sphere, cylinder, axis)
* History of contact lens use and duration
* Prior ocular surgery or trauma, if applicable
* Family history of keratoconus or corneal ectasia
* Use of medications that may influence tear film stability or corneal biomechanics
* Ocular surface disease documentation if present (e.g., dry eye, blepharitis)

Imaging and Diagnostic Data Requirements:

* Availability of at least one valid and complete set of:
* Scheimpflug-based corneal tomography (e.g., Pentacam or equivalent)
* Anterior segment OCT (AS-OCT), if performed
* Epithelial thickness mapping (optional but desirable)
* Corneal biomechanical data (optional)
* Imaging files must be:
* Of adequate quality as judged by the original technician and reviewer
* Free from significant artifacts or motion blur
* Properly labeled by eye (OD/OS) and imaging modality
* Acquired with standard scan protocols

Diagnostic Spectrum Requirements:

* Patients may fall into any of the following diagnostic categories:
* Normal cornea eligible for laser refractive surgery
* Suspect keratoconus or forme fruste keratoconus
* Established keratoconus of any stage (I-IV or ABCD)
* Post-CXL (cross-linking) cornea undergoing follow-up evaluation
* Post-keratoplasty cornea (e.g., DALK, PKP) undergoing diagnostic review
* Patients disqualified from surgery due to abnormal tomography or other contraindications.

Exclusion Criteria:

1. Incomplete or Poor Quality Data:

   * Patients with missing, incomplete, or poor-quality clinical data or corneal imaging that precludes reliable diagnosis by either AI or consultant review.
2. Ocular Comorbidities:

   * Presence of ocular diseases that could confound the diagnosis or interpretation of refractive error or keratoconus, such as advanced glaucoma, active uveitis, significant retinal pathology, or previous corneal transplantation.
3. Severe Systemic Disease Affecting the Eye:

   * Patients with systemic diseases known to affect the cornea or refraction (e.g., connective tissue disorders with corneal involvement) will be excluded to avoid confounding effects.
4. Inability or Refusal to Consent:

   * For prospectively enrolled cases, patients (or guardians, in the case of minors) who are unwilling or unable to provide informed consent will be excluded.
5. Participation in Conflicting Studies:

   * Patients currently enrolled in other interventional studies that could interfere with the diagnostic process or outcomes measured in this study.

Clinical Documentation Exclusions:

* Missing or incomplete visual acuity data.
* Absence of manifest refraction or subjective refraction data.
* Incomplete or conflicting patient history with unresolvable discrepancies.
* Absence of necessary demographic identifiers (e.g., gender, age, laterality of findings).

Imaging and Data Quality Exclusions:

* Imaging datasets with significant artifacts that preclude AI analysis.
* Files missing key parameters (e.g., Belin/Ambrósio D index, Kmax, pachymetry) required for keratoconus classification.
* Inability to determine laterality (OD/OS) for specific scans.
* Scans acquired with outdated or non-standard imaging protocols.
* Mislabeling or duplication of imaging sets across different patients.

Case-Type Exclusions:

* Cases involving active ocular infection or inflammation at the time of evaluation.
* Cases with active herpetic eye disease, corneal ulcer, or epithelial defects interfering with imaging interpretation.
* Prior laser refractive surgery unless explicitly classified and used as part of post-refractive ectasia evaluation.
* Eyes with concurrent advanced retinal pathology that may confound diagnostic interpretation (e.g., macular edema, retinal dystrophies).

Technology-Specific Exclusions:

* Imaging performed using devices not compatible with the AEYE data ingestion framework (e.g., certain older corneal topographers).
* Non-English documentation incompatible with NLP parsing in the General Ophthalmology Agent.

Other Considerations:

* AEYE must be able to process the case within its defined schema. If key data elements are absent or the case causes schema failure, it will be excluded from quantitative analysis but may be reported qualitatively as part of system performance limitations.
* If multiple attempts at AI processing result in non-deterministic or erroneous outputs, such cases will be logged but excluded from primary outcome evaluation.
* Human reviewers (consultant ophthalmologists) must have completed their diagnostic interpretation independently prior to AEYE input; any cases where human opinion was influenced by AI output will be excluded to preserve blinding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes 50 anonymized patient cases collected from a private ophthalmology clinic. Patients were originally evaluated either for refractive surgery-including LASIK or other vision correction procedures-or for suspected or known keratoconus. Each case includes complete clinical documentation and high-quality corneal imaging (e.g., Pentacam, AS-OCT). The study population represents a typical clinical spectrum, including normal eyes, early or forme fruste keratoconus, post-CXL, and post-keratoplasty cases. All data was de-identified and retrospectively analyzed to assess the diagnostic performance of the AEYE system against expert human evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Multi-Agent AI Workflow Compared to Consultant Ophthalmologist | From January 2020 to the anticipated study completion date (including retrospective review of cases from 2020 and prospective enrollment of new cases through 2025)
  The primary outcome is the diagnostic accuracy of the orchestrated multi-agent AI workflow (AEYE) for detecting refractive errors and keratoconus, compared to independent diagnoses made by a consultant ophthalmologist. Accuracy will be assessed by calculating sensitivity, specificity, positive and negative predictive values, and overall concordance between AI and consultant findings. All assessments are blinded, and discrepancies will be adjudicated by a review panel. Both retrospective and prospective cases are included to capture real-world performance over a broad patient population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazem Yassin Clinics, Cairo, Maadi, Egypt

REFERENCES:
- [Background] MedHELM: Holistic Evaluation of Large Language Models for Medical Tasks By: Suhana Bedi, Hejie Cui, Miguel Fuentes, Alyssa Unell, Michael Wornow, Juan M. Banda, Nikesh Kotecha, Timothy Keyes, Yifan Mai, Mert Oez, Hao Qiu, Shrey Jain, Leonardo Schettini, Mehr Kashyap, Jason Alan Fries, Akshay Swaminathan, Philip Chung, Fateme Nateghi, Asad Aali, Ashwin Nayak, Shivam Vedak, Sneha S. Jain, Birju Patel, Oluseyi Fayanju, Shreya Shah, Ethan Goh, Dong-han Yao, Brian Soetikno, Eduardo Reis, Sergios Gatidis, Vasu Divi, Robson Capasso, Rachna Saralkar, Chia-Chun Chiang, Jenelle Jindal, Tho Pham, Faraz Ghoddusi, Steven Lin, Albert S. Chiou, Christy Hong, Mohana Roy, Michael F. Gensheimer, Hinesh Patel, Kevin Schulman, Dev Dash, Danton Char, Lance Downing, Francois Grolleau, Kameron Black, Bethel Mieso, Aydin Zahedivash, Wen-wai Yim, Harshita Sharma, Tony Lee, Hannah Kirsch, Jennifer Lee, Nerissa Ambers, Carlene Lugtu, Aditya Sharma, Bilal Mawji, Alex Alekseyev, Vicky Zhou, Vikas Kakkar, Jarrod Helzer, Anurang Revri, Yair Bannett, Roxana Daneshjou, Jonathan Chen, Emily Alsentzer, Keith Morse, Nirmal Ravi, Nima Aghaeepour, Vanessa Kennedy, Akshay Chaudhari, Thomas Wang, Sanmi Koyejo, Matthew P. Lungren, Eric Horvitz, Percy Liang, Mike Pfeffer, Nigam H. Shah Journal: arxiv arXiv:2505.23802v2 Submitted on 26 May 2025 (v1), last revised 2 Jun 2025
- [Background] Olawade DB, Weerasinghe K, Mathugamage MDDE, Odetayo A, Aderinto N, Teke J, Boussios S. Enhancing Ophthalmic Diagnosis and Treatment with Artificial Intelligence. Medicina (Kaunas). 2025 Feb 28;61(3):433. doi: 10.3390/medicina61030433. PMID 40142244
- [Background] Hubbard DC, Cox P, Redd TK. Assistive applications of artificial intelligence in ophthalmology. Curr Opin Ophthalmol. 2023 May 1;34(3):261-266. doi: 10.1097/ICU.0000000000000939. Epub 2022 Dec 29. PMID 36728651
- See also: Authoritative resource on keratoconus pathophysiology, staging, and management — https://www.aao.org/eye-health/diseases/what-is-keratoconus
- See also: Provides context on refractive surgery evaluation and contraindications — https://americanrefractivesurgerycouncil.org/lasik-candidacy-the-complete-screening-guide/
- See also: Details key imaging device and parameters used in AEYE workflow — https://www.pentacam.com/us/start.html
- See also: Describes the core orchestration framework used to implement AEYE's multi-agent design — https://docs.dify.ai/en/guides/workflow/README